CLINICAL TRIAL: NCT06869902
Title: Is Inhaled Colostrum as Effective as Inhaled Lavender Essential Oil for Pain Control in Neonatal Frenotomy: A Prospective, Randomized Clinical Trial
Brief Title: Use of Inhaled Colostrum to Control Pain in Neonatal Frenotomy and Comparison to Inhaled Lavender Essential Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023/10996
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-09

CONDITIONS: Pain; Ankyloglossia; Neonate
Keywords: ankyloglossia; lavender; colostrum; pain
MeSH Terms: conditions — Pain; Ankyloglossia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A blinded observer assessed pain by means of the Neonatal Infant Pain Scale (NIPS) score, crying duration, and whether there was a change in heart rate (HR) and/or in oxygen saturation (satO2) before and after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender essential oil (No Intervention): Patients were swaddled, were given 1 mL of oral sucrose, and we let them suck for 2 minutes prior to the procedure. We placed a 7 x 7 cm gauze pad with 1 drop (43.75 mg) of 100% pure LEO (Pranarôm España S.L.) 2 cm under their nose for 2 minutes prior to starting the frenotomy and for the duration of the procedure.
- Colostrum (Experimental): Patients were swaddled, were given 1 mL of oral sucrose, and we let them suck for 2 minutes prior to the procedure. We placed a 7 x 7 cm gauze pad with 2 drops of their mother's colostrum 2 cm under their nose for 2 minutes prior to starting the frenotomy and for the duration of the procedure.
  Interventions: Biological: Colostrum

INTERVENTIONS:
Biological: Colostrum — Use of the patient's mother's inhaled colostrum during the frenotomy
  Arms: Colostrum

SUMMARY:
Neonatal pain must be treated because it may have long-term negative effects. Frenotomy (clipping the tongue-tie) is a painful procedure where common strategies to relieve pain (give oral sucrose, let the baby suck, etc) cannot be used because the technique is performed on the tongue. Inhaling lavender essential oil (LEO) helps treat pain during painful procedures such as blood sampling, vaccination, and frenotomy. We aimed to determine whether smelling colostrum had similar effects as inhaled LEO during frenotomies. We conducted a prospective, randomized clinical trial between September 2023 and June 2024 and evaluated babies who underwent a frenotomy. We assessed pain using the NIPS score, heart rate, oxygen saturation, and crying time. After obtaining parental informed consent, we randomized patients into experimental and control groups. In both groups, we performed swaddling, administered oral sucrose, and let the newborn suck for 2 minutes. In the experimental group, we placed a gauze pad with two drops of colostrum, whereas in the control group, we used one drop of LEO 2 cm under the neonate's nose prior to and during the frenotomy.

DETAILED DESCRIPTION:
We conducted a prospective, randomized clinical trial. Our hospital Ethics Committee (CEIm-PSMAR) approved this study (reference code: 2023/10996). Prior to patient enrollment we obtained a signed informed consent from the neonate's parents. This study was conducted according to the ethics code of the Barcelona Medical Association and the principles of the Helsinki-Fortaleza Declaration 2013, at the neonatal unit of a tertiary care hospital in Barcelona (Spain) within an area of influence of approximately 400,000 people, which experiences approximately 1,400 births per year. The target population for this study, and thus, inclusion criteria were healthy full-term neonates born at our center or less than 15 days old referred for a frenotomy, who had ankyloglossia according to the Hazelbaker tool between September 2023 and June 2024. We assess for the presence of ankyloglossia as part of the routine neonatal evaluation using the Hazelbaker tool to evaluate its impact on tongue movement and on breastfeeding. According to the Hazelbaker tool, ankyloglossia exists if appearance scores 8 points or less and/or function scores 11 points or less. We offer a frenotomy to all patients with ankyloglossia. During the study period, if we identified a patient with ankyloglossia, we offered the patient's parents the opportunity to participate in this study.

Patients were enrolled if their parents agreed to and signed a written informed consent. We only included patients who were breastfed, as after randomization we may need to get colostrum. Enrolled patients were randomized into case or control group by simple random sampling using sequentially numbered containers. During the frenotomy the neonate was taken to the neonatal unit and monitored with a pulse-oximeter (COVIDIEN Nellcor Portable SpO2 Patient Monitoring System PM10N, Covidien Ireland Limited, IDA Business & Technology Park, Tullamore, Ireland) before, during and after the procedure. For both groups we swaddled, administered 1 mL of oral sucrose, and let the newborn suck for 2 minutes prior to the procedure. The control group had a 7 x 7 cm gauze pad with 1 drop (43.75 mg) of 100% pure LEO (Pranarôm España S.L.) placed 2 cm under their nose for 2 minutes prior to starting the frenotomy and for the duration of the procedure, whereas the experimental group had a gauze with 2 drops of colostrum of the patient's mother placed in the same way. We used two drops of colostrum but only one of LEO because the odor of colostrum is more subtle than that of LEO, and in our previous studies [32-33] we had used one drop of LEO, and that is how we routinely perform frenotomies. Once the procedure was completed, we removed the gauze pad and recorded vital signs, whether the baby cried or not, the seconds crying lasted, and the NIPS score on a data collection sheet. If a neonate cried, calming techniques such as holding, swaddling, and sucking were employed. A blinded observer assessed pain by means of the Neonatal Infant Pain Scale (NIPS) score (Figure 2) [40], crying duration, and whether there was a change in heart rate (HR) and/or in oxygen saturation (satO2) before and after the procedure.

In a previously published study where we compared performing frenotomies using complementary analgesia or not with inhaled LEO, we observed a mean (SD) crying time of 14.8 vs 24.6 (10.8 vs 27.6) seconds in favor of LEO [32]. In order to detect a difference of 10 seconds in crying time, we calculated that we needed a sample size of 71 patients per group in order to draw conclusions with a CI 95% and a power of 80%. We chose to evaluate pain by means of the increase of HR rather than via the NIPS score because in previous research, we obtained NIPS scores of 1.88-2.92 and 2.02-2.38, and a NIPS score less than 3 indicates no pain. We used the NIPS score to assess whether neonates exhibited pain when using inhaled colostrum instead of LEO.

We recorded demographic (sex, gestational age, birth weight, age in hours at the time of frenotomy) and clinical variables (HR and satO2 before, during, and after the procedure, whether the patient cried or not during the procedure, length of crying time in seconds, presence of side effects during the procedure (apnea, desaturation, others) and highest NIPS score within the first 5 minutes after the procedure). The attending staff were trained to assess the NIPS score before we started recruiting patients. Even though patients were swaddled, it was feasible to feel if they moved their legs or arms. The independent variable was the use of inhaled colostrum or inhaled LEO during frenotomy. The dependent variables were HR and satO2 pre and post procedure, presence of crying and duration, hours of life at the time of the frenotomy, and the NIPS score. The controlled variables were gestational age, sex, and birth weight.

Statistical analysis: Quantitative variables (gestational age, birth weight, age at frenotomy, heart rate pre and post-procedure, increase in heart rate post-procedure, oxygen saturation pre and post-procedure, decrease in oxygen saturation post-procedure, and duration of crying) are described using the mean, standard deviation and range; experimental vs control groups were compared with a Student's t-test. We assessed the equality of variances by using Levene's test and applied the result of the Student's t-test accordingly. Sex, the presence of crying, and adverse effects between the two groups are presented in percentages and compared using Fisher's exact test. Statistical significance was set for a p <0.05. To perform statistical analyses we used STATA version 16.1 (StataCorp, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy full-term neonates born at our center or less than 15 days old referred for a frenotomy, who had ankyloglossia according to the Hazelbaker tool who were breastfed

Exclusion Criteria:

* Denial of the patient's parents to participate

Ages: 1 Hour to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Increase in heart rate | Immediately before the technique and up to 5 minutes after completing it
  Increase in heart rate before and after the procedure
Oxygen saturation | Immediately before the technique and up to 5 minutes after completing it
  Decrease in oxygen saturation before and after the procedure
NIPS score | Immediately before the technique and up to 5 minutes after completing it
  Assessment of the highest Neonatal Infant Pain Scale (NIPS) score

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Maya-Enero, PhD, MD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request

REFERENCES:
- [Background] Marlier L, Gaugler C, Messer J. Olfactory stimulation prevents apnea in premature newborns. Pediatrics. 2005 Jan;115(1):83-8. doi: 10.1542/peds.2004-0865. PMID 15629985
- [Background] Vaziri F, Khosropoor M, Hidari M, Pourahmad S, Morshed Behbahani B, Saki F. The Effect of Aromatherapy by Lavender Oil on Infant Vaccination Pain: a Double Blind Randomized Controlled Trial. J Caring Sci. 2019 Mar 1;8(1):17-21. doi: 10.15171/jcs.2019.003. eCollection 2019 Mar. PMID 30915309
- [Background] Cetinkaya B, Basbakkal Z. The effectiveness of aromatherapy massage using lavender oil as a treatment for infantile colic. Int J Nurs Pract. 2012 Apr;18(2):164-9. doi: 10.1111/j.1440-172X.2012.02015.x. PMID 22435980
- [Background] Burns E, Blamey C, Ersser SJ, Lloyd AJ, Barnetson L. The use of aromatherapy in intrapartum midwifery practice an observational study. Complement Ther Nurs Midwifery. 2000 Feb;6(1):33-4. doi: 10.1054/ctnm.1999.0901. PMID 11033651
- [Background] Habanananda T. Non-pharmacological pain relief in labour. J Med Assoc Thai. 2004 Oct;87 Suppl 3:S194-202. PMID 21213523
- [Background] Lopez V, Nielsen B, Solas M, Ramirez MJ, Jager AK. Exploring Pharmacological Mechanisms of Lavender (Lavandula angustifolia) Essential Oil on Central Nervous System Targets. Front Pharmacol. 2017 May 19;8:280. doi: 10.3389/fphar.2017.00280. eCollection 2017. PMID 28579958
- [Background] Akcan E, Polat S. Comparative Effect of the Smells of Amniotic Fluid, Breast Milk, and Lavender on Newborns' Pain During Heel Lance. Breastfeed Med. 2016 Aug;11(6):309-314. doi: 10.1089/bfm.2015.0174. Epub 2016 Jun 17. PMID 27315487
- [Background] Goubet N, Rattaz C, Pierrat V, Bullinger A, Lequien P. Olfactory experience mediates response to pain in preterm newborns. Dev Psychobiol. 2003 Mar;42(2):171-80. doi: 10.1002/dev.10085. PMID 12555281
- [Background] Harrison D, Larocque C, Bueno M, Stokes Y, Turner L, Hutton B, Stevens B. Sweet Solutions to Reduce Procedural Pain in Neonates: A Meta-analysis. Pediatrics. 2017 Jan;139(1):e20160955. doi: 10.1542/peds.2016-0955. Epub 2016 Dec 16. PMID 27986905
- [Background] Blass EM, Miller LW. Effects of colostrum in newborn humans: dissociation between analgesic and cardiac effects. J Dev Behav Pediatr. 2001 Dec;22(6):385-90. doi: 10.1097/00004703-200112000-00006. PMID 11773803
- [Background] Bellieni CV, Buonocore G, Nenci A, Franci N, Cordelli DM, Bagnoli F. Sensorial saturation: an effective analgesic tool for heel-prick in preterm infants: a prospective randomized trial. Biol Neonate. 2001 Jul;80(1):15-8. doi: 10.1159/000047113. PMID 11474143
- [Background] Bellieni CV, Bagnoli F, Perrone S, Nenci A, Cordelli DM, Fusi M, Ceccarelli S, Buonocore G. Effect of multisensory stimulation on analgesia in term neonates: a randomized controlled trial. Pediatr Res. 2002 Apr;51(4):460-3. doi: 10.1203/00006450-200204000-00010. PMID 11919330
- [Background] Carbajal R, Veerapen S, Couderc S, Jugie M, Ville Y. Analgesic effect of breast feeding in term neonates: randomised controlled trial. BMJ. 2003 Jan 4;326(7379):13. doi: 10.1136/bmj.326.7379.13. PMID 12511452
- [Background] Ludington-Hoe SM, Hosseini R, Torowicz DL. Skin-to-skin contact (Kangaroo Care) analgesia for preterm infant heel stick. AACN Clin Issues. 2005 Jul-Sep;16(3):373-87. doi: 10.1097/00044067-200507000-00010. PMID 16082239
- [Background] Johnston CC, Stevens B, Pinelli J, Gibbins S, Filion F, Jack A, Steele S, Boyer K, Veilleux A. Kangaroo care is effective in diminishing pain response in preterm neonates. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1084-8. doi: 10.1001/archpedi.157.11.1084. PMID 14609899
- [Background] Gray L, Watt L, Blass EM. Skin-to-skin contact is analgesic in healthy newborns. Pediatrics. 2000 Jan;105(1):e14. doi: 10.1542/peds.105.1.e14. PMID 10617751
- [Background] Blass EM, Hoffmeyer LB. Sucrose as an analgesic for newborn infants. Pediatrics. 1991 Feb;87(2):215-8. PMID 1987534
- [Background] Stevens B, Yamada J, Ohlsson A, Haliburton S, Shorkey A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2016 Jul 16;7(7):CD001069. doi: 10.1002/14651858.CD001069.pub5. PMID 27420164
- [Background] Blass EM, Ciaramitaro V. A new look at some old mechanisms in human newborns: taste and tactile determinants of state, affect, and action. Monogr Soc Res Child Dev. 1994;59(1):I-V, 1-81. PMID 8047076
- [Background] Field T, Goldson E. Pacifying effects of nonnutritive sucking on term and preterm neonates during heelstick procedures. Pediatrics. 1984 Dec;74(6):1012-5. PMID 6504620
- [Background] Fitri SYR, Wardhani V, Rakhmawati W, Pahria T, Hendrawati S. Culturally Based Practice in Neonatal Procedural Pain Management: A Mini Review. Front Pediatr. 2020 Sep 3;8:540. doi: 10.3389/fped.2020.00540. eCollection 2020. PMID 33014934
- [Background] Razaghi N, Aemmi SZ, Sadat Hoseini AS, Boskabadi H, Mohebbi T, Ramezani M. The effectiveness of familiar olfactory stimulation with lavender scent and glucose on the pain of blood sampling in term neonates: A randomized controlled clinical trial. Complement Ther Med. 2020 Mar;49:102289. doi: 10.1016/j.ctim.2019.102289. Epub 2019 Dec 26. PMID 32147068
- [Background] Franck LS, Lawhon G. Environmental and behavioral strategies to prevent and manage neonatal pain. Semin Perinatol. 1998 Oct;22(5):434-43. doi: 10.1016/s0146-0005(98)80059-1. PMID 9820568
- [Background] Simons SH, van Dijk M, Anand KS, Roofthooft D, van Lingen RA, Tibboel D. Do we still hurt newborn babies? A prospective study of procedural pain and analgesia in neonates. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1058-64. doi: 10.1001/archpedi.157.11.1058. PMID 14609893
- [Background] Carbajal R, Rousset A, Danan C, Coquery S, Nolent P, Ducrocq S, Saizou C, Lapillonne A, Granier M, Durand P, Lenclen R, Coursol A, Hubert P, de Saint Blanquat L, Boelle PY, Annequin D, Cimerman P, Anand KJ, Breart G. Epidemiology and treatment of painful procedures in neonates in intensive care units. JAMA. 2008 Jul 2;300(1):60-70. doi: 10.1001/jama.300.1.60. PMID 18594041
- [Background] Mitchell A, Boss BJ. Adverse effects of pain on the nervous systems of newborns and young children: a review of the literature. J Neurosci Nurs. 2002 Oct;34(5):228-36. doi: 10.1097/01376517-200210000-00002. PMID 12391738
- [Background] Johnston C. Pain control in infants and young children. Pain Res Manag. 2011 Sep-Oct;16(5):320. doi: 10.1155/2011/505039. No abstract available. PMID 22059203
- [Result] Field T, Field T, Cullen C, Largie S, Diego M, Schanberg S, Kuhn C. Lavender bath oil reduces stress and crying and enhances sleep in very young infants. Early Hum Dev. 2008 Jun;84(6):399-401. doi: 10.1016/j.earlhumdev.2007.10.008. Epub 2007 Nov 28. PMID 18053656
- [Result] Rattaz C, Goubet N, Bullinger A. The calming effect of a familiar odor on full-term newborns. J Dev Behav Pediatr. 2005 Apr;26(2):86-92. doi: 10.1097/00004703-200504000-00003. PMID 15827459
- [Result] Yilmaz F, Arikan D. The effects of various interventions to newborns on pain and duration of crying. J Clin Nurs. 2011 Apr;20(7-8):1008-17. doi: 10.1111/j.1365-2702.2010.03356.x. Epub 2010 Nov 5. PMID 21054600
- [Result] Neshat H, Jebreili M, Seyyedrasouli A, Ghojazade M, Hosseini MB, Hamishehkar H. Effects of Breast Milk and Vanilla Odors on Premature Neonate's Heart Rate and Blood Oxygen Saturation During and After Venipuncture. Pediatr Neonatol. 2016 Jun;57(3):225-31. doi: 10.1016/j.pedneo.2015.09.004. Epub 2015 Oct 20. PMID 26560183
- [Result] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Result] Karadede H, Mutlu B. The Effect of Swaddling and Oropharyngeal Colostrum During Endotracheal Suctioning on Procedural Pain and Comfort in Premature Neonates: A Randomized Controlled Trial. Adv Neonatal Care. 2024 Oct 1;24(5):466-474. doi: 10.1097/ANC.0000000000001190. Epub 2024 Aug 27. PMID 39141691
- [Result] Nishitani S, Miyamura T, Tagawa M, Sumi M, Takase R, Doi H, Moriuchi H, Shinohara K. The calming effect of a maternal breast milk odor on the human newborn infant. Neurosci Res. 2009 Jan;63(1):66-71. doi: 10.1016/j.neures.2008.10.007. Epub 2008 Nov 1. PMID 19010360
- [Result] Maya-Enero S, Fabregas-Mitjans M, Llufriu-Marques RM, Candel-Pau J, Garcia-Garcia J, Lopez-Vilchez MA. Comparison of the analgesic effect of inhaled lavender vs vanilla essential oil for neonatal frenotomy: a randomized clinical trial (NCT04867824). Eur J Pediatr. 2022 Nov;181(11):3923-3929. doi: 10.1007/s00431-022-04608-3. Epub 2022 Sep 8. PMID 36076107
- [Result] Maya-Enero S, Fabregas-Mitjans M, Llufriu-Marques RM, Candel-Pau J, Garcia-Garcia J, Lopez-Vilchez MA. Analgesic effect of inhaled lavender essential oil for frenotomy in healthy neonates: a randomized clinical trial. World J Pediatr. 2022 Jun;18(6):398-403. doi: 10.1007/s12519-022-00531-7. Epub 2022 Apr 4. PMID 35377106
- [Result] Slater R, Cornelissen L, Fabrizi L, Patten D, Yoxen J, Worley A, Boyd S, Meek J, Fitzgerald M. Oral sucrose as an analgesic drug for procedural pain in newborn infants: a randomised controlled trial. Lancet. 2010 Oct 9;376(9748):1225-32. doi: 10.1016/S0140-6736(10)61303-7. PMID 20817247
- [Result] Ors R, Ozek E, Baysoy G, Cebeci D, Bilgen H, Turkuner M, Basaran M. Comparison of sucrose and human milk on pain response in newborns. Eur J Pediatr. 1999 Jan;158(1):63-6. doi: 10.1007/s004310051011. PMID 9950311
- [Result] Goubet N, Strasbaugh K, Chesney J. Familiarity breeds content? Soothing effect of a familiar odor on full-term newborns. J Dev Behav Pediatr. 2007 Jun;28(3):189-94. doi: 10.1097/dbp.0b013e31802d0b8d. PMID 17565285
- [Result] Leng HY, Zheng XL, Zhang XH, He HY, Tu GF, Fu Q, Shi SN, Yan L. Combined non-pharmacological interventions for newborn pain relief in two degrees of pain procedures: A randomized clinical trial. Eur J Pain. 2016 Jul;20(6):989-97. doi: 10.1002/ejp.824. Epub 2015 Dec 18. PMID 26685099
- [Result] Walter-Nicolet E, Annequin D, Biran V, Mitanchez D, Tourniaire B. Pain management in newborns: from prevention to treatment. Paediatr Drugs. 2010 Dec 1;12(6):353-65. doi: 10.2165/11318900-000000000-00000. PMID 21028915

DOCUMENTS (3):
  • Study Protocol (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT06869902/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT06869902/SAP_001.pdf
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT06869902/ICF_002.pdf